CLINICAL TRIAL: NCT06985615
Title: A Multi-center, Parallel Cohort, Open Label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of HDM1002 in Subjects With Normal Hepatic Function and Hepatic Impairment.
Brief Title: A Study of HDM1002 in Subjects With And Without Varying Degrees Of Hepatic Impairement
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDM1002-109
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: HDM1002

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subjects Without Hepatic Impairment (Experimental)
  Interventions: Drug: Single dose of HDM1002 on Day 1
- Subjects With Mild Hepatic Impairment (Experimental)
  Interventions: Drug: Single dose of HDM1002 on Day 1
- Subjects With Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: Single dose of HDM1002 on Day 1
- Subjects With Severe Hepatic Impairment (Experimental)
  Interventions: Drug: Single dose of HDM1002 on Day 1

INTERVENTIONS:
Drug: Single dose of HDM1002 on Day 1 — Single dose of HDM1002 will be administered on Day 1

SUMMARY:
The current study is proposed to evaluate whether there is any clinically meaningful effect of hepatic impairment on the plasma Pharmacokinetic (PK) of HDM1002

ELIGIBILITY:
Inclusion Criteria:

1. Age and Sex: Chinese subjects aged 18-70 years (inclusive) at screening, regardless of gender. The normal hepatic function group and hepatic impairment group must be age-matched within ±10 years, with gender matching as close as possible (±1 subject per gender).
2. Body Weight and Body Mass Index (BMI): At screening, male subjects must weigh ≥50.0 kg, and female subjects ≥40.0 kg, with a BMI ranging from 19.0 to 32.0 kg/m² (inclusive).The normal hepatic function group and hepatic impairment group must be weight-matched within ±10 kg.

Exclusion Criteria:

1. History or family history of medullary thyroid carcinoma, thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2; or serum calcitonin ≥50 ng/L at screening.
2. History of chronic pancreatitis or an episode of acute pancreatitis within 3 months prior to signing the informed consent form (ICF).
3. History of acute gallbladder disease within 3 months prior to signing the ICF.
4. History of Malignancy: Diagnosis of any malignancy within 5 years prior to ICF signing (except basal cell carcinoma treated with curative intent and deemed cured).
5. Severe Systemic Diseases: History of severe cardiovascular, neuropsychiatric, gastrointestinal, respiratory, urinary, endocrine, or other systemic diseases (e.g., acute myocardial infarction, severe depression, gastric ulcer, uremia) within 1 year prior to ICF signing.
6. Conditions Affecting Drug Pharmacokinetics: Presence of dysphagia or any condition that, on the investigator's judgment, may impact drug absorption, distribution, metabolism, or excretion (e.g., active inflammatory bowel disease, gastrectomy, intestinal resection) at screening.
7. Severe Hypoglycemia: Episode of severe hypoglycemia within 3 months prior to screening.
8. Allergy or Intolerance: History of allergic diseases (e.g., asthma, urticaria, eczematous dermatitis) or known intolerance/allergy to glucagon-like peptide-1 receptor (GLP-1R) agonists.
9. Hepatic Function Normal Group Exclusions:a) History of chronic liver disease, including hepatitis, hepatitis B, or hepatitis C, or positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (anti-HCV) at screening.b) Positive Treponema pallidum antibody.c) Use of any medication within 28 days or 5 elimination half-lives (whichever is longer) prior to the first study drug administration.
10. Hepatic Impairment Group Exclusions:a) Hepatocellular carcinoma, hepatorenal syndrome, or limited life expectancy (defined as <1 year for the hepatic impairment cohort).b) Cirrhosis complications (e.g., gastrointestinal bleeding, severe hypoglycemia) within 3 months prior to screening.c) Use of any medication within 7 days or 5 half-lives (whichever is longer) prior to the first study drug administration that may affect HDM1002 pharmacokinetics (PK).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Predose (0 hours), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post dose.
  Maximum observed plasma of HDM1002 concentration.
Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) | Predose (0 hours), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post dose.
  Area under the plasma HDM1002 concentration-time profile from time 0 extrapolated to infinite time.
Area Under the Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) | Predose (0 hours), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post dose.
  Area under the plasma HDM1002 concentration-time profile from time 0 extrapolated to the time of the last quantifiable concentration.
Fraction of Unbound Drug in Plasma (fu) | Predose (0 hours), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post dose.
  fu = Cu/C (where Cu represents unbound concentration and C represents total concentration).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China